CLINICAL TRIAL: NCT00761280
Title: Efficacy and Safety of AP 12009 in Adult Patients With Recurrent or Refractory Anaplastic Astrocytoma or Secondary Glioblastoma as Compared to Standard Chemotherapy Treatment: A Randomized, Actively Controlled, Open Label Clinical Phase III Study.
Brief Title: Efficacy and Safety of AP 12009 in Patients With Recurrent or Refractory Anaplastic Astrocytoma or Secondary Glioblastoma
Acronym: SAPPHIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit the projected patient number. All analyses are descriptive, only.
Sponsor: Isarna Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 12009-G005
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Anaplastic Astrocytoma; Glioblastoma
Keywords: Anaplastic astrocytoma; Glioblastoma; Antisense; Cancer; Transforming Growth Factor beta 2; Targeted therapy; Brain tumor; Glioma; Central Nervous System (CNS); Convection Enhanced Delivery (CED); Intratumoral administration
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Neoplasms; Brain Neoplasms; Glioma | interventions — Trabedersen; Temozolomide; Drug Delivery Systems; Carmustine; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trabedersen 10 µM (Experimental): 10 µM trabedersen (AP 12009), intratumoral infusion, every other week, 11 cycles, maximum 21 weeks
  Interventions: Drug: trabedersen; Device: Drug delivery system for administration of AP 12009; Procedure: Placement of Drug Delivery System
- Chemotherapy (Active Comparator): temozolomide: capsules, up to 200 mg/sqm/day, 5 days per cycle, up to 26 cycles; carmustine: i.v. administration, up to 200 mg/sqm/day, 1 day per cycle, up to 8 cycles; lomustine: capsules, 110 mg/sqm/day, 1 day per cycle, up to 8 cycles. Only 1 of these 3 drugs/interventions is administered per patient in the comparator arm.
  Interventions: Drug: temozolomide; Drug: carmustine; Drug: lomustine

INTERVENTIONS:
Drug: trabedersen
  Other Names: AP 12009
  Arms: trabedersen 10 µM
Drug: temozolomide
  Other Names: Temodar; Temodal; TMZ
  Arms: Chemotherapy
Device: Drug delivery system for administration of AP 12009 — Drug delivery system for Convection Enhanced Delivery consists of a portable pump (Pegasus vario or Pega vario) with drug reservoir (Pega Bag) and infusion line (Pega Line). Main implanted parts are the port access system (PORT-A-CATH) and the intratumoral catheter (Medtronic ventricular catheter).
  Arms: trabedersen 10 µM
Procedure: Placement of Drug Delivery System — Surgery for placement of intratumoral catheter and subcutaneous port access system as per routine clinical practice. Stereotactical catheter placement controlled by CT.
  Arms: trabedersen 10 µM
Drug: carmustine
  Other Names: BCNU; BiCNU; Carmubris
  Arms: Chemotherapy
Drug: lomustine
  Other Names: CCNU; CeeNU
  Arms: Chemotherapy

SUMMARY:
In this multinational Phase III study the efficacy and safety of 10 µM AP 12009 is compared to standard chemotherapy (temozolomide or BCNU or CCNU) in adult patients with confirmed recurrent or refractory anaplastic astrocytoma (WHO grade III) or secondary glioblastoma (WHO grade IV).

DETAILED DESCRIPTION:
The purpose of this study is to compare the safety and efficacy of the 10 µM concentration of AP 12009 and standard chemotherapy (temozolomide, BCNU, CCNU) in adult patients with recurrent or refractory anaplastic astrocytoma (AA, WHO grade III) or secondary glioblastoma (GBM, WHO grade IV). AP 12009 (trabedersen) is a phosphorothioate antisense oligodeoxynucleotide specific for the mRNA of human Transforming Growth Factor beta 2 (TGF-beta-2), which is applied intratumorally. The growth factor TGF-beta plays a key role in malignant progression of various tumors by inducing proliferation, invasion, metastasis, angiogenesis, and escape from immunosurveillance. In patients with high-grade glioma, the TGF-beta-2 overexpression is associated with disease stage, clinical prognosis, and the immunodeficient state of the patients. Main objective of the study is to determine survival (rate) and tumor response.

Important note: Due to early trial termination, resulting in limited data availability, all analyses remain descriptive by nature, only. No conclusive endpoint analysis can be performed.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent prior to any study-related procedure.
* The patient is at least 18 years of age and equal to or below 70 years.
* The patient has a present diagnosis of AA or secondary GBM.
* The patient has a measurable lesion (> 1 ccm in volume, central MRI review).
* The lesion (or sum of lesions) does not exceed 50 ccm in volume (central MRI review).
* The tumor is localized supratentorially (central MRI review).
* All patients have recurrent or refractory disease, i.e. disease has progressed after prior surgery and radiotherapy at any time of the disease course or stage. Secondary GBM patients have progressed after a previous diagnosis of A and/or AA.
* The patient has not received more than one chemotherapy regimen. Radiation with concomitant chemotherapy, followed by adjuvant chemotherapy, is considered as one chemotherapy regimen.
* The patient is eligible for chemotherapy.
* The patient is on a maximum dose of 4 mg/day dexamethasone or equivalent doses for other corticosteroids, which has been stable or decreasing for at least 3 weeks prior to Screening.
* The patient is male or a non-pregnant, non-lactating female.
* Females of childbearing potential must have a negative beta-HCG pregnancy test at Screening.
* Females of childbearing potential and males must practice strict birth control.
* The patient must have recovered from acute toxicity caused by any previous therapy.
* The patient has a life expectancy of at least 3 months.
* The patient has a Karnofsky Performance Status of at least 70%.
* The patient shows adequate organ functions as assessed by the following screening laboratory values:

  1. Adequate renal function determined by serum creatinine and urea < 2 times the upper limit of normal
  2. Adequate liver function with ALT, AST and AP < 3 times the upper limit of normal, and bilirubin < 2.5 mg/dL
  3. INR < 1.5 and aPTT < 1.5 x ULN
  4. Hemoglobin > 9 g/dL
  5. Platelet count > 100 x 10E9/L
  6. WBC > 3 x 10E9/L
  7. ANC > 1.5 x 10E9/L (or WBC > 3.0 x 10E9/L)

Exclusion Criteria:

* Patient unable or not willing to comply with the protocol regulations.
* The investigator deems it necessary to surgically (re-)resect the present tumor (NOTE: the patient might still be eligible for randomization at a later timepoint).
* Tumor surgery, tumor debulking, or other neurosurgery within 3 months prior to randomization. If a ≤48-hour routine post-surgery MRI (in accordance with study specifications) qualifies the patient for study participation, the patient can be randomized 30 ± 7 days post-surgery.
* Radiotherapy or stereotactic (gamma knife) radiosurgery within 3 months prior to randomization.
* Prior interstitial brachytherapy of the brain with permanent implants. Prior interstitial brachytherapy of the brain with removable implants within 3 months prior to randomization.
* Chemotherapy, hormone therapy, or any other therapy with established or suggested anti-tumor effects within 4 weeks (nitrosoureas: 6 weeks) prior to randomization.
* Prior anti-TGF-beta 2 targeted therapy.
* Screening MRI shows a mass effect caused by the tumor defined as significant compression of the ventricular system and/or a midline shift (≥ 3 mm, central MRI review). Compression of the ventricular system and/or a midline shift ≥ 3 mm only due to the presence of (a) cyst(s) or scarring processes does not exclude an individual from the study.
* Participation in another clinical study with another investigational medicinal product within 30 days prior to randomization.
* History of a second independent malignant disorder within 5 years, except for carcinoma in situ of the cervix and basal cell carcinoma.
* Presence of poorly controlled seizures.
* Clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure, unstable angina, or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomization.
* Known HIV, HBV or HCV infection.
* Acute viral, bacterial, or fungal infection.
* Acute medical problems that may be considered to become an unacceptable risk, or any conditions, which might be contraindications for starting study treatment.
* Presence of high risk for pulmonary toxicities, defined as:

  1. Lung function: vital capacity ≤ 70%
  2. Status following sequential or concomitant thoracic irradiation
  3. Increased risk for a pulmonary toxicity induced by BCNU (Carmustine) or CCNU (Lomustine). Risk factors include smoking, presence of a respiratory condition, pre-existing radiographic pulmonary abnormalities, exposure to agents that cause lung damage.
* History of allergies to reagents used in this study, history of celiac disease.
* Drug abuse or extensive use of alcohol.
* Clinically relevant psychiatric disorders / legal incapacity or a limited legal capacity.
* Concomitant treatment with yellow fever vaccine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Del Maestro, MD, PhD, Study Chair — Montreal Neurological Institute and Hospital
Locations (68):
- United States (3):
  - NJ Neuroscience Institute; JFK Medical Center, Edison, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - University of Rochester Medical Center, Rochester, New York
- Argentina (3):
  - Hospital Británico, Buenos Aires
  - FLENI, Buenos Aires
  - Sanatorio Allende, Córdoba
- Austria (2):
  - Universitätsklinik Innsbruck, Abteilung für Neurologie, Innsbruck
  - AKH Wien, Klinik für Neurochirurgie, Vienna
- Brazil (6):
  - Hospital de Câncer de Barretos, Barretos / SP
  - Centro Goiano de Oncologia (CGO), Goiânia
  - Hospital Sao Vicente de Paulo, Passo Fundo
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital do Servidor Público Estadual, São Paulo
- Canada (3):
  - ECOGENE-21 Centre d'études cliniques, Chicoutimi, Quebec
  - Foothills Medical Centre, Calgary
  - Montreal Neurological Institute and Hospital, Montreal
- La Timone University Hospital, Marseille, France
- Germany (10):
  - Klinik und Poliklinik für Neurochirurgie, Frankfurt/M.
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Neurochirurgische Klinik an der Universität Ulm am Bezirkskrankenhaus Günzburg, Günzburg
  - Universitätklinikum Hamburg-Eppendorf, Klinik für Neurochirurgie, Hamburg
  - Medizinische Hochschule Hannover Neurochirurgische Klinik, Hanover
  - Universitätsklinik Heidelberg Neurologische Klinik, Heidelberg
  - Universitätsklinikum Leipzig, Neurochirurgische Klinik, Leipzig
  - Otto-von-Guericke-Universität, Klinik für Neurochirurgie, Magdeburg
  - Klinik und Poliklinik für Neurochirurgie, Münster
  - Klinik und Poliklinik für Neurologie, Regensburg
- Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Hungary
- India (12):
  - Manipal Hospital & Manipal Institute for Neurological Disorders, Bangalore
  - NIMHANS, Bangalore
  - BGS Global Hospital, Bangalore
  - Postgraduate Institute of Medical Education & Research (PGIMER), Chandigarh
  - Apollo Speciality Hospitals, Chennai
  - Care Hospitals, Hyderabaad
  - Amrita Institute of Medical Sciences Research Center, Kochi
  - AMRI Hospitals, Kolkata
  - SGPGI of Medical Sciences, Lucknow
  - Advanced Centre for Treatment Research and Education in Cancer (ACTREC), Mumbai
  - All India Institute of Medical Sciences (AIIMS), New Delhi
  - SCTIMST, Dept. of Neurosurgery, Thiruvananthapuram
- Mexico (3):
  - Hospital San Javier, Guadalajara
  - Hospital General de Mexico, Mexico City
  - Medica Sur, Mexico City
- Poland (6):
  - Wojskowy Szpital Kliniczny, Klinika Neurochirurgii, Bydgoszcz
  - Akademickie Centrum Kliniczne, Gdansk
  - SP ZOZ Uniwersytecki Szpital Kliniczny nr 1, Klinika Neurochirurgii, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Klinika Neurochirurgii i Neurochirurgii Dziecięcej, Lublin
  - Kliniczny Oddzial Neurochirurgii SUM w Sosnowcu Wojewódzki Szpital Specjalistyczny nr 5, Sosnowiec
  - Centrum Onkologii - Instytut Im. Marii Sklodowskiej-Curie, Warsaw
- Russia (5):
  - Chelyabinsk City Hospital #3; Department of Neurosurgery, Chelyabinsk
  - State Institution Russian Oncology Research Center N.N. Blokhin, Moscow
  - Russian Scientific Research Neurosurgical Institute A.L. Polenov, Saint Petersburg
  - Military Medical Academy, Neurosurgery Dept, Saint Petersburg
  - Samara Region Clinical Hospital M.I. Kalinin, Samara
- South Korea (3):
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Kangnam St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital de Cruces, Barakaldo
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Doce de Octubre, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
- United Kingdom (2):
  - Edinburgh Centre for Neuro-Oncology, Western General Hospital, Edinburgh
  - The National Hospital for Neurology and Neurosurgery, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Temozolomide: capsules, up to 200 mg/sqm/day, 5 days per cycle, up to 26 cycles.
  OR carmustine: i.v. administration, up to 200 mg/sqm/day, 1 day per cycle, up to 8 cycles;
  OR lomustine: capsules, 110 mg/sqm/day, 1 day per cycle, up to 8 cycles.
  Only 1 of these 3 drugs/interventions is administered per patient in the comparator arm.
Period: Randomization to First Dose
Arm/Group | Trabedersen 10 µM | Chemotherapy
Started | 14 | 13
Catheter Surgery | 13 (Safety population) | 0 (Not applicable to control group)
First Dose of Study Drug / Chemotherapy | 12 | 11 (Safety population)
Completed | 12 | 11
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor decision | 1 | 0
Not completed — Other | 1 | 0
Period: First Dose to End of Study
Arm/Group | Trabedersen 10 µM | Chemotherapy
Started | 12 | 11
Completed | 0 (Study was discontinued early due to the inability to recruit a sufficient number of participants.) | 0 (Study was discontinued early due to the inability to recruit a sufficient number of participants.)
Not Completed | 12 | 11
Not completed — End of trial | 5 | 5
Not completed — Progressive disease | 5 | 3
Not completed — Sponsor decision | 1 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population includes all participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabedersen 10 µM | Chemotherapy | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.72) | 40.8 (11.63) | 39.5 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 10 | 18
  Black | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Hispanic or Latino | 0 | 1 | 1
  American Indian or Native Alaskan | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Study was discontinued early because of the inability to recruit a sufficient number of suitable participants within the planned recruitment period, therefore not all planned sites recruited participants. Only those regions that recruited at least one participant are listed.
  participants
    Spain | 1 | 1 | 2
    Austria | 0 | 1 | 1
    Russian Federation | 4 | 4 | 8
    India | 6 | 2 | 8
    Mexico | 0 | 1 | 1
    Canada | 0 | 1 | 1
    Germany | 1 | 2 | 3
    Israel | 0 | 1 | 1
    Poland | 2 | 0 | 2
Height (cm) (Descriptive analysis, only) [Mean (Standard Deviation); unit: cm] — Height is missing for one participant in the Chemotherapy group.
  cm | 172.57 (9.913) | 170.29 (10.019) | 171.52 (9.829)
Weight (kg) (Descriptive analysis, only) [Mean (Standard Deviation); unit: kg] — Weight is missing for one participant in the Chemotherapy group.
  kg | 75.34 (17.265) | 71.62 (14.213) | 73.62 (15.731)
Diagnosis of Anaplastic Astrocytoma (AA) World Health Organization (WHO) Grade III [Number; unit: participants] — Twenty-six participants were diagnosed with Anaplastic Astrocytoma, and one participant was diagnosed with Secondary Glioblastoma Multiforme.
  participants
    Refractory | 3 | 2 | 5
    Recurrent | 11 | 10 | 21
Time of first diagnosis of AA WHO Grade III (years) (Descriptive analysis, only) [Mean (Standard Deviation); unit: years] — Time of first diagnosis (in years before study entry) is available for all 14 participants in the Trabedersen group and 11 participants in the chemotherapy group.
  years | 1.71 (1.110) | 1.81 (1.194) | 1.75 (1.124)
Diagnosis of other brain tumor prior to diagnosis of Anaplastic Astrocytoma WHO Grade III [Number; unit: participants] — Twenty-six participants were diagnosed with Anaplastic Astrocytoma, and one participant was diagnosed with Secondary Glioblastoma Multiforme.
  participants
    AA WHO Grade I | 0 | 0 | 0
    AA WHO Grade II | 1 | 0 | 1
    Not diagnosed with Other Brain Tumor | 12 | 12 | 24
    Other diagnosis | 1 | 0 | 1
Diagnosis of Secondary Glioblastoma Multiforme (GBM) (WHO Grade IV) [Number; unit: participants] | 0 | 1 | 1
Time to first diagnosis of Secondary GBM (years) (Descriptive analysis, only) [Mean (Standard Deviation); unit: years] — Time of first diagnosis (in years before study entry) of Secondary Glioblastoma Multiforme. One participant in the Chemotherapy group was diagnosed with Secondary Glioblastoma Multiforme (GBM); all other participants were diagnosed with Anaplastic Astrocytoma (AA).
  years | NA (NA) — No participants in this group were diagnosed with Secondary Glioblastoma Multiforme. | 0.03 (NA) — One participant in this group was diagnosed with Secondary Glioblastoma Multiforme. | 0.03 (NA) — One participant in this group was diagnosed with Secondary Glioblastoma Multiforme.
Previous diagnosis of Astrocytoma or AA before diagnosis of Secondary Glioblastoma Multiforme [Number; unit: participants]
  Previous diagnosis of Astrocytoma | 0 | 0 | 0
  Previous diagnosis of Anaplastic Astrocytoma | 0 | 1 | 1
One or more Prior Surgical Treatments [Number; unit: participants]
  Yes | 14 | 12 | 26
  No | 0 | 1 | 1
One or more Prior Radiotherapy Regimens [Number; unit: participants] | 14 | 13 | 27
One or more Prior Chemotherapy [Number; unit: participants]
  Yes | 10 | 9 | 19
  No | 4 | 4 | 8
One or more Prior Immunotherapy [Number; unit: participants]
  Yes | 1 | 1 | 2
  No | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at 24 Months in the Intent-to-treat Population - Percentage of Participants (Descriptive Analysis, Only)
Description: Survival rate was defined as the proportion of participants known to be alive at 24 months from randomization. If a participant's status was unknown and there was no follow-up information available, they were categorized as 'Died' for the purposes of the analysis.
Time Frame: 24 months
Population: The Intent-to-treat population includes all participants randomized. Early study discontinuation with site closures led to a high proportion of participants being censored or lost to follow-up in the initial analysis. Additional survival data were collected in a post-hoc fashion under a protocol amendment. These data are presented.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
percentage of participants | 28.6 [11.7 to 54.6] | 15.4 [4.3 to 42.2]

2. Secondary Outcome: Survival Rate at 12, 18, and 21 Months in the Intent-to-treat Population - Percentage of Participants (Descriptive Analysis, Only)
Description: Survival rate was defined as the proportion of participants known to be alive at each time-point from randomization. Participants with unknown or missing status were considered treatment failures, i.e., assumed to be dead.
Time Frame: 12, 18, and 21 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
percentage of participants
  Survival rates at 12 months | 57.1 [32.6 to 78.6] | 53.8 [29.1 to 76.8]
  Survival rates at 18 months | 42.9 [21.4 to 67.4] | 38.5 [17.7 to 64.5]
  Survival rates at 21 months | 35.7 [16.3 to 61.2] | 23.1 [8.2 to 50.3]

3. Secondary Outcome: Survival at 12, 18, and 21 Months in the Intent-to-treat Population - Number of Participants
Description: Survival status was assessed at each time-point from randomization. Participants with unknown or missing status were considered treatment failures, i.e., assumed to be dead. The category "Lost to follow-up" for each time-point includes participants who were alive at the last data collection point but did not yet have enough follow-up time to reach the time point.
Time Frame: 12, 18, and 21 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
participants
  Alive at 12 months | 8 | 7
  Died at 12 months | 5 | 1
  Lost to follow-up at 12 months | 1 | 5
  Alive at 18 months | 6 | 5
  Died at 18 months | 7 | 3
  Lost to follow-up at 18 months | 1 | 5
  Alive at 21 months | 5 | 3
  Died at 21 months | 7 | 5
  Lost to follow-up at 21 months | 2 | 5

4. Secondary Outcome: Median Overall Survival (Days) From Randomization in the Intent-to-treat Population (Descriptive Analysis, Only)
Description: Median overall survival was defined as the date of randomization to the date of death. If a participant's status was unknown and there was no follow-up information available, they were categorized as 'Died' for the purposes of the analysis. Analysis was by Kaplan-Meier estimation.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
days | 458.0 [193.0 to NA] — The upper limit of the 95% confidence interval could not be calculated because of insufficient data. | 584.5 [426.0 to NA] — The upper limit of the 95% confidence interval could not be calculated because of insufficient data.

5. Secondary Outcome: Response Category by Independent Review in the Intent-to-treat Population - Number of Participants
Description: Tumor response was classified based on the (neuro-)radiologist's evaluation according to the Macdonald Response Criteria for bidimensionally measurable disease as outlined below:
  * Complete Response (CR): Disappearance of all enhancing tumor on consecutive MRI scans at least 1 month apart, off steroids, neurologically stable or improved.
  * Partial Response (PR): ≥50% reduction in size of enhancing tumor on consecutive MRI scans at least 1 month apart, steroids stable or reduced, neurologically stable or improved.
  * Progressive Disease (PD): ≥25% increase in size of enhancing tumor or any new tumor on MRI scans, steroids stable or increased, neurologically worse.
  * Stable Disease (SD): all other situations.
  Two qualified neuro-radiologists reviewed scans at each MRI time point, with adjudication of discrepancies by a third reviewer. Their findings and clinical information were independently reviewed by a neuro-oncologist, who made the assessment of overall response.
Time Frame: Up to 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Number; unit: participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 1
  Stable Disease (SD) | 2 | 6
  Progressive Disease (PD) | 7 | 1
  Unknown | 1 | 3
  Missing | 2 | 2

6. Secondary Outcome: Overall Response Rate (CR+PR) by Independent Review in the Intent-to-treat Population - Percentage of Participants (Descriptive Analysis, Only)
Description: Overall response rate was the proportion of participants with a best response of Complete Response (CR) or Partial Response (PR) observed from the start of treatment until disease progression.
Time Frame: Up to 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
percentage of participants | 14.3 [4.0 to 39.9] | 7.7 [1.4 to 33.3]

7. Secondary Outcome: Tumor Control Rate (CR+PR+SD) by Independent Review in the Intent-to-treat Population - Percentage of Participants (Descriptive Analysis, Only)
Description: Tumor control rate was defined as the proportion of participants assessed as having Complete Response (CR), Partial Response (PR), or Stable Disease (SD). Participants with unknown or missing response were treated as non-responders.
Time Frame: Up to 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
percentage of participants | 28.6 [11.7 to 54.6] | 53.8 [29.1 to 76.8]

8. Primary Outcome: Survival at 24 Months in the Intent-to-treat Population - Number of Participants
Description: Survival status was assessed at 24 months from randomization. Participants with unknown or missing status were considered treatment failures, i.e., assumed to be dead. The category "Lost to / insufficient follow-up" includes participants who were alive at last data collection point but did not yet have enough follow-up time to reach the 24 month time point.
Time Frame: 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
participants
  Alive | 4 | 2
  Died | 7 | 5
  Lost to/insufficient follow-up | 3 | 6

9. Secondary Outcome: Median Duration of Response (Days) by Independent Review (Descriptive Analysis, Only)
Description: Duration of response was defined as the time from the first documentation of confirmed response (Complete Response, CR, or Partial Response, PR) to the first signs of Progressive Disease (PD), as assessed by the study neuro-oncologist. Median Duration of Response was calculated by Kaplan-Meier estimate.
  Censoring rules were:
  * at the date of randomization -- participants without baseline assessments, or for those with no post-baseline timor assessments who were discontinued for other than progressive disease or death.
  * at the date of last tumor assessment -- discontinuation other than PD or death, or if a new treatment was started prior to disease progression
  * at the date of death or last tumor assessment -- death or PD after one missed tumor assessment
  * at the date of last tumor assessment -- death or PD after more than one missed tumor assessment
  * at the date of last tumor assessment -- participants on ongoing treatment at data cut-off
Time Frame: Up to 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
days | NA [NA to NA] — Due to early discontinuation of study, an insufficient number of patients reached this endpoint for estimation. | NA [NA to NA] — Due to early discontinuation of study, an insufficient number of patients reached this endpoint for estimation.

10. Secondary Outcome: Disease Progression at 10, 12, 14, 16, 18, 21, and 24 Months by Independent Review in the Intent-to-treat Population - Number of Participants
Description: Tumor response was classified based on the (neuro-)radiologist's evaluation:
  * Complete Response (CR): Disappearance of all enhancing tumor on consecutive MRI scans at least 1 month apart, off steroids, neurologically stable or improved.
  * Partial Response (PR): ≥50% reduction in size of enhancing tumor on consecutive MRI scans at least 1 month apart, steroids stable or reduced, neurologically stable or improved.
  * Progressive Disease (PD): ≥25% increase in size of enhancing tumor or any new tumor on MRI scans, steroids stable or increased, neurologically worse.
  * Stable Disease (SD): all other situations.
  Based on clinical and imaging data, an independent neuro-oncologist made the final assessment of "Progressed" versus "Not Progressed". Participants who had MRI assessment results missing or unknown were "UNK or missing", and were treated as "Progressed" for the purposes of the calculation.
Time Frame: 10, 12, 14, 16, 18, 21, and 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Number; unit: participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
participants
  Progressed at 10 months | 7 | 5
  Not progressed at 10 months | 3 | 0
  Status unknown / missing at 10 months | 4 | 7
  Lost to follow-up at 10 months | 0 | 1
  Progressed at 12 months | 7 | 5
  Not progressed at 12 months | 2 | 0
  Status unknown / missing at 12 months | 5 | 7
  Lost to follow-up at 12 months | 0 | 1
  Progressed at 14 months | 7 | 5
  Not progressed at 14 months | 2 | 0
  Status unknown / missing at 14 months | 5 | 7
  Lost to follow-up at 14 months | 0 | 1
  Progressed at 16 months | 7 | 5
  Not progressed at 16 months | 2 | 0
  Status unknown / missing at 16 months | 5 | 7
  Lost to follow-up at 16 months | 0 | 1
  Progressed at 18 months | 7 | 5
  Not progressed at 18 months | 2 | 0
  Status unknown / missing at 18 months | 5 | 7
  Lost to follow-up at 18 months | 0 | 1
  Progressed at 21 months | 7 | 5
  Not progressed at 21 months | 1 | 0
  Status unknown / missing at 21 months | 6 | 7
  Lost to follow-up at 21 months | 0 | 1
  Progressed at 24 months | 7 | 5
  Not progressed at 24 months | 1 | 0
  Status unknown / missing at 24 months | 6 | 7
  Lost to follow-up at 24 months | 0 | 1

11. Secondary Outcome: Disease Progression Rate at 10, 12, 14, 16, 18, 21, and 24 Months by Independent Review in the Intent-to-treat Population - Percentage of Participants (Descriptive Analysis, Only)
Description: as for outcome 10
Time Frame: 10, 12, 14, 16, 18, 21 and 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
percentage of participants
  Progression rate at 10 months | 78.6 [52.4 to 92.4] | 100.0 [77.2 to 100.0]
  Progression rate at 12 months | 85.7 [60.1 to 96.0] | 100.0 [77.2 to 100.0]
  Progression rate at 14 months | 85.7 [60.1 to 96.0] | 100.0 [77.2 to 100.0]
  Progression rate at 16 months | 85.7 [60.1 to 96.0] | 100.0 [77.2 to 100.0]
  Progression rate at 18 months | 85.7 [60.1 to 96.0] | 100.0 [77.2 to 100.0]
  Progression rate at 21 months | 92.9 [68.5 to 98.7] | 100.0 [77.2 to 100.0]
  Progression rate at 24 months | 92.9 [68.5 to 98.7] | 100.0 [77.2 to 100.0]

12. Secondary Outcome: Median Time to Progression (Days) by Independent Review for the Intent-to-treat Population (Descriptive Analysis, Only)
Description: Time to progression was calculated from the date of randomization to the date of the first documented tumor progression. Participants who did not progress or died were censored at the last tumor assessment date or the date of start of a new anti-tumor treatment or death.
Time Frame: Up to 24 months
Population: The Intent-to-treat population includes all participants randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Trabedersen 10 µM | Chemotherapy
Number analyzed (Participants) | 14 | 13
days | 57.0 [57.0 to NA] — The upper limit of the 95% confidence interval was not calculable because of insufficient data. | 153.5 [65.0 to 209.0]

ADVERSE EVENTS:
Time Frame: Safety monitoring (including adverse events) started from the signature of the informed consent and continued until 28 days after the last administration of study drug, up to 24 months.
Description: Only treatment-emergent adverse events are listed, defined as any AE whose onset occurred or intensity worsened after undertaking the first study procedure or first dose of study drug (whichever occurred first) but less than 28 days after medication/procedures had stopped. Adverse events (including lab tests) were assessed at study visits.
Arm/Group | Trabedersen 10 µM | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 6/13 | 0/11
Other Adverse Events (participants affected / at risk) | 12/13 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabedersen 10 µM (N=13) | Chemotherapy (N=11)
Grand mal convulsion (Nervous system disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Meningitis (Infections and infestations) | 2 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neurosurgery (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trabedersen 10 µM (N=13) | Chemotherapy (N=11)
Headache (Nervous system disorders) | 7 (7) | 2 (2)
Partial seizures (Nervous system disorders) | 4 (4) | 0 (0)
Brain oedema (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Facial palsy (Nervous system disorders) | 2 (2) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0)
Acquired epileptic aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0)
Device occlusion (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Administration site reaction (General disorders) | 0 (0) | 1 (1)
Device alarm issue (General disorders) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Neutrophil count (Investigations) | 0 (0) | 2 (2)
White blood cell count (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
CSF protein increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 1 (1)
Pseudomonas test positive (Investigations) | 1 (1) | 0 (0)
Staphylococcus test postivie (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meningitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Hippus (Eye disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Varicose veins (Vascular disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Neurosurgery (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination of the study leading to recruitment of 27 of 180 planned subjects and incomplete collection of data. Survival results are based on post-study collection of additional survival data under a protocol amendment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and Sponsor both have publication / presentation privileges. Investigator abstracts or publications had to be reviewed and approved by the Sponsor prior to submission or presentation. The Clinic/Investigator agrees to delete information or defer publication or presentation, if (i) publication would hinder or delay the development of the investigational product or (ii) necessary to permit the filing of any desired patent applications by the Sponsor.